CLINICAL TRIAL: NCT01116765
Title: Impact of Early Oral Stimulation on Reducing Cardiorespiratory Events and Transition to Oral Feeding in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2009-A01191-56; 2009-27 (Other: 2009-27)
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Preterm Infants
Keywords: preterm infants born between 26 to 29 weeks of gestation age.

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- experimental group (Experimental): Infants in the experimental group receive an oral stimulation program consisting of stimulation of the oral structures during 10 consecutive days
  Interventions: Other: stimulation of the oral structure
- control group (Other): Infant in the control group receive no stimulation only non nutritive sucking during feeding
  Interventions: Other: no stimulation of the oral structure

INTERVENTIONS:
Other: no stimulation of the oral structure
  Arms: control group
Other: stimulation of the oral structure
  Arms: experimental group

SUMMARY:
To assess whether an oral stimulation program, before the introduction of oral feeding, enhances the cardiorespiratory manifestations (episodes of oxygen désaturations, and/or apnea- bradycardia), and the oral feeding performance, in preterm infants born between 26 to 29 weeks of gestation age.

DETAILED DESCRIPTION:
Preterm infant were randomized into an experimental or an control group. Infants in the experimental group receive an oral stimulation program consisting of stimulation of the oral structures during 10 consecutive days. Infant in the control group receive no stimulation only non nutritive sucking during feeding. Both were administered twice per day, during 20 minutes, 48 hours after discontinuation of nasal continuous positive air pressure. A long term evaluation of oral feeding difficulties and neuromotor development are organized.

ELIGIBILITY:
Inclusion Criteria:

* Children whose born term is included between 26 and 29SA past and whose postnatal age is lower or more equal in 33SA past, at the time of the inclusion.
* Term of certain child (calculated according to the date of the last rules and\or a premature obstetric echography).
* Children devoid of neurological pathology making him(it) clinically unstable (echography transfontanellar and\or intellectual MRI, electroencephalogram normal, either, intraventricular bleeding of rank 1 and 2 of Papile [40], or, intellectual abnormalities in the MRI of type(chap) 1 - 4 according to the classification of modified Paneth [41]. (Annex X)
* Children devoid of infectious pathology making him(it) clinically unstable (Protein C-reactive lower than 7).
* In case of ebb gastroenteritis - esophageal symptomatic ( RGO): the child will be treated(handled), by oral route, by location + thickening +/-prokinetic +/-inhibitor pumps in proton.
* According to a protocol of service, all the premature babies of less than 32.

Exclusion Criteria:

* Born Child > 29 limited companies.
* Child not included at the postnatal age of 33 past(over) LIMITED COMPANIES.
* Child presenting a genic syndrome, an evolutionary neurological disease, a pathology malformative.
* Child presenting a bleeding intraventricular of rank 3-4 [ 40 ], intellectual abnormalities in the MRI of type(chap) 5 and 6 according to the classification of modified Paneth [ 41 ], an ulcer-necrotizing entérocolitis.
* Child among whom both relatives(parents) or legal representatives refused that their child participates in the study.

Ages: 29 Weeks to 33 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2010-05-01 (Actual); Primary Completion 2014-02-24 (Actual); Study Completion 2023-04-13 (Actual)

PRIMARY OUTCOMES:
the cardiorespiratory manifestations | 2 years
  to assess whether an oral stimulation program, before the introduction of oral feeding, enhances the cardiorespiratory manifestations

SECONDARY OUTCOMES:
the oral feeding performance | 2 years
  the oral feeding performance

CONTACTS AND LOCATIONS:
Overall Officials: MURIEL BUSUTIL, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France